CLINICAL TRIAL: NCT04337424
Title: Evaluation of Quickly Diagnostic Saliva Tests for SARS-CoV-2
Acronym: EasyCoV
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: societe SkillCell - 97198 Jarry (Unknown); CNRS Alcediag UMR9005 - societe Sys2Diag - 34184 Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0170
Record Dates: First submitted 2020-04-05; First posted 2020-04-07 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV-2
Keywords: Diagnosis test; Salivary sampling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary sampling (1 to 2 ml of salivary)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with active infection test to SARS-COV2: Sampling of saliva (1 to 2 ml)
  Interventions: Diagnostic Test: Sampling salivary
- Convalescent participants for SARS-COV2: Sampling of saliva (1 to 2 ml)
  Interventions: Diagnostic Test: Sampling salivary
- Participants cured to SARS-COV2: Sampling of saliva (1 to 2 ml)
  Interventions: Diagnostic Test: Sampling salivary
- Participants with negative test to SARS-COV2: Sampling of saliva (1 to 2 ml)
  Interventions: Diagnostic Test: Sampling salivary

INTERVENTIONS:
Diagnostic Test: Sampling salivary — Collection of 1 to 2 ml of saliva

SUMMARY:
Coronavirus disease 2019 or COVID-19 is a highly contagious infectious disease. Symptoms of the disease are non-specific (fever, cough, dyspnea and fatigue), common with many seasonal viruses, which complicates the diagnosis. For mild forms, which represent the vast majority of cases, hospitalization is not necessary and treatment is symptomatic. However in more severe cases, hospitalization is required and sometimes even admission to an intensive care unit.

Several diagnostic tests are already available, but they require, in all cases, the intervention of qualified health personnel to carry out the sample, which includes a risk of contagion and an expensive and time-consuming laboratory analysis and reagents. These tests are therefore not very suitable for massive screenings.

We want to evaluate the performance of a detection test performed on a salivary sample in the diagnosis of SARS-CoV-2. This test will be non-invasive, performed without any analytical device and will restore its qualitative result "infected versus non-infected" in less than 1 hour (30min objective).

DETAILED DESCRIPTION:
Study taking place at the Montpellier University Hospital, comparing a salivary sample group with active infection (participants) for SARS-COV2 with a salavary sample tested negative (cured, convalescent and negative) for SARS-COV2 (healthcare workers ,participants)

ELIGIBILITY:
Inclusion Criteria:

- Control subjects (COV2- group): Participants ( Healthcare staff, patients and DRIVE participants) negative for SARS-CoV-2

- Infected subjects (COV2 + group): Patients diagnosed positive for SARS-CoV-2 hospital staff known to be positive and coming to do a control PCR DRIVE participants.

Exclusion Criteria:

* Eligibility Criteria:

Inclusion Criteria:

- Control subjects (COV2- group): Healthcare staff presumed and diagnosed negative for SARS-CoV-2

- Infected subjects (COV2 + group): Patients diagnosed positive for SARS-CoV-2 hospital staff known to be positive and coming to do a control PCR

Exclusion Criteria:

* Not affiliated with a French Social Security Systemscheme or equivalent system
* Persons deprived of their liberty, adult protected under guardianship or vulnerable persons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The samples size is 90 samples with active infection to SARS-COV2 and at least 90 with no active infection
Sampling Method: Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Specific detection of SARS-CoV-2 specific RNA | 1 day
  Detection by the LAMP method is to be corroborated with the reference method, RT-PCR on the same salivary sample. Only one sample is taken per subject participating in the study. The sample is divided into two aliquots which will be analyzed by LAMP and RT-PCR

SECONDARY OUTCOMES:
Analytical sensitivity of the LAMP test. | 1 day
  This test developed by SYS2DIAG / SKILLCELL must be able to detect a minimum viral load equivalent to that of the standard method on the same salivary sample.
The correlation between the measurement of the assayed viral load (CT value) by the standard method and by the LAMP developed by SYS2DIAG / SKILLCELL. | 1 day
  A correlation between the viral loads measured on the same sample by RT-PCR and by LAMP will be carried out.
Evaluation of the use of saliva samples compared to nasopharyngeal samples | 1 day
  The RT-PCR results on these 2 types of samples and the LAMP results for the saliva samples will be compared with the patient diagnosis to assess the feasibility and performance of the saliva samples for the molecular diagnosis of SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: REYNES Jacques, PU PH, Principal Investigator — Montpellier Hospital
Locations (1):
- UCH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No